CLINICAL TRIAL: NCT05803551
Title: A Phase II Randomized, Double Blind, Placebo-Controlled Study Evaluating the Effects of Ketamine Infusions in Clinically Depressed ICU Patients
Brief Title: A Study of Ketamine Infusions to Treat Clinically-depressed ICU Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Devang Sanghavi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-004767
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Experimental): Adult patients who have been in the Mayo Clinic Florida ICU for one week with moderate or severe depression will receive intravenous (IV) ketamine
  Interventions: Drug: Ketamine Hydrochloride
- Placebo Group (Placebo Comparator): Adult patients who have been in the Mayo Clinic Florida ICU for one week with moderate or severe depression will receive intravenous (IV) placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Intravenous 0.5 mg/kg infusions of ketamine for three consecutive days, 24 hours apart, with no more than 1mg/kg or 60 mg/day regardless of body weight
  Other Names: Ketalar
  Arms: Ketamine Group
Drug: Placebo — Intravenous 0.9% saline infusions for three consecutive days.
  Arms: Placebo Group

SUMMARY:
The purpose of this research is to study the effects of intravenous ketamine infusions for the treatment of patients with depressive symptoms in intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Has been in the Mayo Clinic Florida ICU for the past 1 week.
* PHQ-9 score of 10 or higher.
* One of the following diagnoses: acute myocardial infarction; acute renal failure; chronic obstructive pulmonary disease (COPD); congestive heart failure; end-stage liver disease; patients requiring intra-aortic balloon pump (IABP) therapy or continuous renal replacement therapy (CRRT); post-bone marrow transplant; acute Hypoxemic Respiratory Failure; acute or chronic hypoxemic respiratory failure; pre- or post- lung, liver or heart transplant or surgical overflows (such as abdominal aortic aneurysm, thoracotomy or tracheostomy).

Exclusion Criteria:

* Poor vital sign stability hypoxia: O2 < 95%, hypotension: SBP < 90 hypertension: SBP > 180.
* Heart rate: < 50 or > 120, or Respiratory Rate: < 10 or > 30.
* Altered mental status.
* Patient is unwilling to participate or provide informed consent.
* Any allergy to ketamine or diphenhydramine.
* Patient is female of child-bearing age and unwilling to provide urine or blood for HCG analysis.
* Pregnant or breastfeeding.
* Presence of intracranial mass or vascular lesion.
* Presence of a history of psychosis or hallucinations (as assessed by electronic chart review).
* Weight greater than 115 kg or less than 45kg.
* History of increased intracranial pressure/hypertensive hydrocephalus or increased intraocular pressure.
* Patient is acutely psychotic.
* Provider feels that patient currently or likely will require chemical and/or physical restraints.
* History of prolonged QT-interval.
* Current treatment includes any medication known to affect the N-methyl-D-aspartate receptor system (e.g., lamotrigine, acamprosate, memantine, riluzole, or lithium).
* Patient in withdrawal from substance abuse or who have used hallucinogens (including cannabis) in the last month for any indication, as determined by the clinical interview and urine drug screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | Baseline, 7 days after third infusion
  Evaluated by Patient Health Questionnaire-9 (PHQ-9) used to assess degree of depression severity rating symptoms on a scale of 0=not at all, 3=nearly everyday. Higher score indicates greater depression severity.
Clinically significant improvement of depressive symptoms | 24 hours after initial infusion
  Number of subjects to show clinically significant improvement in depressive symptoms, defined as a reduction in the PHQ-9 of 5 points or more.
Clinically significant improvement of depressive symptoms | 24 hours after third infusion
  Number of subjects to show clinically significant improvement in depressive symptoms, defined as a reduction in the PHQ-9 of 5 points or more.
Clinically significant improvement of depressive symptoms | 14 days after third infusion
  Number of subjects to show clinically significant improvement in depressive symptoms, defined as a reduction in the PHQ-9 of 5 points or more.

CONTACTS AND LOCATIONS:
Overall Officials: Devang Sanghavi, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials